CLINICAL TRIAL: NCT02291393
Title: The Role of High Density Surface Cardiac Electrographic Mapping in the Diagnosis of Arrhythmogenic Right Ventricular Cardiomyopathy :A Pilot Study
Brief Title: The Role of High Density Surface ECG in the Diagnosis of Arrhythmogenic Right Ventricular Cardiomyopathy (ARVC)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Leeds Teaching Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CD12/10936; 12/YH/0346 (Other: Research Ethics Committee)
Record Dates: First submitted 2014-11-11; First posted 2014-11-14 (Estimated); Last update posted 2015-05-19 (Estimated); Status verified 2015-05

CONDITIONS: Arrhythmogenic Right Ventricular Cardiomyopathy
MeSH Terms: conditions — Arrhythmogenic Right Ventricular Dysplasia

ARMS (2):
- Patient (Other): Patients with previously confirmed Arrhythmogenic Right Ventricular Cardiomyopathy (ARVC)
  Interventions: Device: 80 lead ECG
- Healthy volunteers (Other): Aged and gender matched healthy controls.
  Interventions: Device: 80 lead ECG

INTERVENTIONS:
Device: 80 lead ECG

SUMMARY:
The diagnosis of Arrhythmogenic right ventricular cardiomyopathy can be difficult. The 80 lead ECG may increase the specificity and sensitivity in diagnosing this potentially life threatening inherited cardiac condition. This pilot would form the basis of a much larger clinical trial to test the utility of this novel diagnostic tool.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a confirmed diagnosis of arrhythmogenic right ventricular cardiomyopathy who are being followed up in the cardiology clinic

Exclusion Criteria:

* Inability to consent
* Pacing dependent patients
* Other concomitant cardiag disease e.g. coronary artery disease
* Atrial fibrillation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-08; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
QRS wave dispersion in an ECG | 5 minutes
  The difference in QRS wave dispersion between the right and left ventricular leads